CLINICAL TRIAL: NCT05659472
Title: The Effect of Combination Mindfulness Spiritual-Based Cognitive Therapy Plus Hypnosis on Levels of Cortisol, Serotonin, and Depression Degree in HIV Patients With Depression
Brief Title: The Effect of Combination Mindfulness Spiritual-Based Cognitive Therapy Plus Hypnosis in HIV Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Technology Institute of Cendekia Utama Kudus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eny Pujiati
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Hypnosis; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: The intervention group was given a combination of mindfulness spiritual-based cognitive therapy (MSBCT) plus hypnosis and the control group was given mindfulness-based cognitive therapy (MBCT).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The process of randomization to determine the respondents into the intervention and control groups without being known by the researchers and respondents.
  Assessment of cortisol, serotonin, and depression levels was not known by researchers, respondents, and care providers and was only known by the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group = Combination mindfulness spiritual-based cognitive therapy plus hypnosis (Experimental): Given to the intervention group with a frequency of once a week for eight weeks. Each session for 120 minutes or 2 hours with a set of MSBCT intervention packages resulting from modified mindfulness-based cognitive therapy with using the mindfulness concept of Kabat Zinn and the five-step model of mindfulness developed by Vidyamala Burch.
  Interventions: Behavioral: Combination mindfulness spiritual-based cognitive therapy plus hypnosis
- Control group = Mindfulness-based cognitive therapy (Experimental): Given to the control group with a frequency of once a week for eight weeks. Each session is 90 minutes or 1.5 hours with a set of MBCT intervention packages developed by Teasdale, 2014
  Interventions: Behavioral: Mindfulness-based cognitive therapy

INTERVENTIONS:
Behavioral: Combination mindfulness spiritual-based cognitive therapy plus hypnosis — The intervention was divided into eight components in eight sessions, namely (1) psychoeducation and intention, (2) awareness of breathing mindfulness, (3) body scan, (4) comfort training through daily activity/comfort exercises, (5) self-compassion / having a great soul with acceptance, gratitude, and sincerity, (6) planning happiness through independent healthy behavior targets, (7) independent healthy behavior (8) independent healthy behavior evaluation. Each therapeutic component of each session is further divided into three sub-components, namely psychoeducation, training, and hypnosis.
  Other Names: Combination MSBCT plus hypnosis
  Arms: Intervention group = Combination mindfulness spiritual-based cognitive therapy plus hypnosis
Behavioral: Mindfulness-based cognitive therapy — The program curriculum consists of the automatic pilot; living in our heads; gathering the scattered mind; recognizing aversion; allowing and letting be; thoughts as thoughts; kindness in action; maintaining and extending new learning.
  Other Names: MBCT
  Arms: Control group = Mindfulness-based cognitive therapy

SUMMARY:
HIV/AIDS patients are at risk for depression, a multifactorial disorder with signs and symptoms that affect the cognitive, affective, behavioral, and somatic areas. This study used Randomized Controlled Clinical Trials (RCT).

Main hypothesis: A combination of spiritual awareness-based cognitive therapy (MSBCT) plus hypnotic interventions can reduce depression degree scores by reducing cortisol levels and increasing serotonin levels in HIV patients with depression.

Small hypothesis

1. There was a decrease in cortisol levels after being given the MSBCT plus hypnosis combination intervention in HIV patients with depression;
2. There was an increase in serotonin levels after being given the MSBCT plus hypnosis combination intervention in HIV patients with depression;
3. There was a decrease in depression degree scores after being given the MSBCT plus hypnosis combination intervention in HIV patients with depression;
4. There was a higher reduction in cortisol levels in the intervention group compared to the control group in HIV patients with depression;
5. There was a higher increase in serotonin levels in the intervention group compared to the control group in HIV patients with depression;
6. There was a higher reduction in scores degree of depression in the intervention group compared to the control group in HIV patients with depression;
7. Decreased cortisol levels and increased serotonin levels affect depression degree scores in HIV patients with depression;
8. MSBCT plus hypnosis combination intervention is a factor that can affect depression degree scores reduction in HIV patients with depression;

DETAILED DESCRIPTION:
HIV/AIDS patients are at risk for depression. Evidence shows that depression in HIV/AIDS patients is two to four times higher than in the general population. The prevalence of depression in HIV/AIDS patients varies from 5% to 79% worldwide while the prevalence of depression in Indonesia in 2018 was 21.8% where women (22.3%) had a higher depression rate than men (21,4%). Cases of depression in HIV/AIDS patients are estimated to have a frequency of up to 60% of the total existing cases of depression.

Depressive disorders are caused by biopsychosocial factors and neurotransmitter interactions that affect pathophysiology in a complex manner. The monoaminergic neurotransmitters that play the most role in depression are serotonin (5-HT), norepinephrine (NE), and dopamine (DA). In people with maladaptive PLHIV, cortisol levels in the blood will increase thereby inhibiting cellular and humoral immune responses. This condition causes apoptosis not to occur so that the virus proliferates and spreads rapidly. The progressive effect of HIV/AIDS can infect the central nervous system thereby disrupting the balance of neurotransmitters, accelerating viral replication, and suppressing the immune response so that it can shorten the period of HIV without symptoms. This condition, if not handled properly can reduce the quality of life, weaken physical function and therapeutic effects, as well as higher medical co-morbidities including suicidal behavior.

Although the prevalence is quite high, the efficacy of depression therapy is currently not satisfactory. Less than 50% of depressed patients respond to standard therapy and 70% relapse. Psychopharmacology, psychotherapy, and a combination of the two are effective for treating depression and preventing the recurrence of depression. Psychopharmacological therapy has a shorter impact than psychotherapy. Even today, many people switch from medical therapy to psychotherapy because of the high medical costs and the side effects of pharmacological therapy. Therefore, equipping HIV/AIDS patients with coping strategies to manage physiological and psychological problems is integral to part of providing comprehensive care to HIV/AIDS patients.

The results of the meta-analysis reported that mindfulness-based therapy was effective in reducing symptoms of stress, anxiety, and depression. There is empirical evidence supporting the effectiveness of MBCT in reducing rates of depression and improving the quality of life in chronic disease patients. However, the study results have not been consistent. Two resources that are widely used by patients with mental and physical illnesses are psychotherapy and religion/spirituality. The results of a meta-analysis of 46 spiritual intervention studies reported that patients with spiritually integrated psychotherapy showed positive improvement compared to patients treated only with psychotherapy. On this basis, researchers are trying to develop MBCT psychotherapy with spiritually integrated MBCT, namely a mindfulness-based intervention that integrates Islamic spiritual values (gratitude, patience, pleasure, sincerity, and trustworthiness) with aspects of cognitive behavioral therapy (CBT) and focuses on current conditions, emphasizes acceptance of thoughts, emotions, and behavior by improving thought processes, controlling emotions, and bodily sensations in order to develop self-capacity effectively in dealing with problems.

Positive self-capacity development can occur and be effective when having the basic principles of positive life in the subconscious mind. One way to explore the subconscious mind can be done with hypnosis. Hypnosis is a method of giving suggestions by penetrating the critical factors of the conscious mind into the subconscious mind. Hypnosis has also been shown to be significant in reducing stress, anxiety, and depression scores. Even hypnosis plays a significant role as the first step in treating depression. This makes researchers try to develop a spiritually integrated MBCT psychotherapy combined with hypnosis.

Formulation of the problem Can a combination intervention of mindfulness spiritual-based cognitive therapy (MSBCT) plus hypnosis reduce depression degree scores by reducing cortisol levels and increasing serotonin levels in HIV patients with depression?

Research purposes The research aims to prove that a combination intervention of mindfulness spiritual-based cognitive therapy (MSBCT) plus hypnosis can reduce depression degree scores by decreasing cortisol levels and increasing serotonin levels in HIV patients with depression.

Research hypothesis A combination intervention of mindfulness spiritual-based cognitive therapy (MSBCT) plus hypnosis can reduce depression degree scores by reducing cortisol levels and increasing serotonin levels in HIV patients with depression.

Benefits of research results Provide scientific information about the effects interventions of a combination of mindfulness spiritual-based cognitive therapy (MSBCT) plus hypnosis in reducing cortisol levels, increasing serotonin levels, and reducing the scores degree of depression in HIV patients with depression;

Research methods A randomized controlled trial (RCT). The sampling used a consecutive sampling method, namely a sampling technique based on inclusion and exclusion criteria for selecting predetermined subjects, within a certain period of time until the number of research subjects was fulfilled. After selecting the subjects, the randomization process was carried out using random allocation. The enumerator determined that each group consisted of 31 subjects in the intervention group and 31 subjects in the control group. Randomization used the simple randomization technique, namely by making 62 envelopes, each with 31 envelopes bearing the combination of MSBCT plus Hypnosis and 31 envelopes bearing the words MBCT. All envelopes were randomized and each subject who met the research criteria received one envelope chosen by the enumerator without the researcher and the subject knowing about it. If the envelope taken contains the writing of the MSBCT plus Hypnosis combination then the subject is included in the intervention group sample and the one containing the MBCT writing is included in the control group sample. The intervention was given once a week for 8 weeks. The assessment was carried out 2 times pre and post-intervention by assessing cortisol levels, serotonin levels, and depression degree scores in the control and intervention groups. Statistical tests used the Independent T-test if the data were normally distributed, the Mann Whitney U Test if the data were not normally distributed, and to see the effect of the intervention using a linear regression test.

ELIGIBILITY:
Inclusion Criteria:

1. HIV patients with mild-moderate depression;
2. Receiving ARV therapy;
3. Islam;
4. Aged 18-60 years;
5. Not taking steroid and serotonin medications;
6. Willing to sign the informed consent;

Exclusion Criteria:

1. Having a history of immune disorders or allergies;
2. Currently undergoing hormonal or corticosteroid therapy;
3. Patients who used herbal medicine 2 weeks before the study;
4. Patients with psychiatric comorbidities and emergency conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Decreased serum cortisol levels | Before intervention, and 8 weeks after intervention
  Serum cortisol levels were measured using the ELISA kit catalog method number CO103S in the GAKI laboratory, Faculty of Medicine, Diponegoro University - Semarang - Indonesia
Increased serum serotonin levels | Before intervention, and 8 weeks after intervention
  Serum serotonin levels were measured using the ELISA kit catalog method number E - EL-H0033 in the GAKI laboratory, Faculty of Medicine, Diponegoro University - Semarang - Indonesia
Decreased degree scores of depression | Before intervention, and 8 weeks after intervention
  Depression degree scores were measured using the Beck Depression Inventory (BDI) II

CONTACTS AND LOCATIONS:
Overall Officials: Eny Pujiati, M.Kes, Principal Investigator — Health Technology Institute of Cendekia Utama Kudus - Middle Java - Indonesia
Locations (1):
- Eny Pujiati, Kudus, Middle Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
I did'd have a plan share the date

REFERENCES:
- [Result] Asangbeh SL, Sobngwi JL, Ekali GL, Eyoum C, Msellati P. Predictors of depression among patients on art in a rural health district in North West Cameroon. AIDS Care. 2016;28(2):205-8. doi: 10.1080/09540121.2015.1074654. Epub 2015 Aug 19. PMID 26288104
- [Result] Bernard C, Dabis F, de Rekeneire N. Prevalence and factors associated with depression in people living with HIV in sub-Saharan Africa: A systematic review and meta-analysis. PLoS One. 2017 Aug 4;12(8):e0181960. doi: 10.1371/journal.pone.0181960. eCollection 2017. PMID 28783739
- [Result] Dejman M, Ardakani HM, Malekafzali B, Moradi G, Gouya MM, Shushtari ZJ, Alinaghi SA, Mohraz M. Psychological, Social, and Familial Problems of People Living with HIV/AIDS in Iran: A Qualitative Study. Int J Prev Med. 2015 Dec 23;6:126. doi: 10.4103/2008-7802.172540. eCollection 2015. PMID 26900440
- [Result] Nanni MG, Caruso R, Mitchell AJ, Meggiolaro E, Grassi L. Depression in HIV infected patients: a review. Curr Psychiatry Rep. 2015 Jan;17(1):530. doi: 10.1007/s11920-014-0530-4. PMID 25413636
- [Result] Feuillet P, Lert F, Tron L, Aubriere C, Spire B, Dray-Spira R; Agence Nationale de Recherche sur le Sida et les Hepatites Virales (ANRS)-VIH: Enquete sur les personnes atteintes (Vespa2) Study Group. Prevalence of and factors associated with depression among people living with HIV in France. HIV Med. 2017 Jul;18(6):383-394. doi: 10.1111/hiv.12438. Epub 2016 Sep 14. PMID 27625202
- [Result] Wang T, Fu H, Kaminga AC, Li Z, Guo G, Chen L, Li Q. Prevalence of depression or depressive symptoms among people living with HIV/AIDS in China: a systematic review and meta-analysis. BMC Psychiatry. 2018 May 31;18(1):160. doi: 10.1186/s12888-018-1741-8. PMID 29855289
- [Result] Uthman OA, Magidson JF, Safren SA, Nachega JB. Depression and adherence to antiretroviral therapy in low-, middle- and high-income countries: a systematic review and meta-analysis. Curr HIV/AIDS Rep. 2014 Sep;11(3):291-307. doi: 10.1007/s11904-014-0220-1. PMID 25038748
- [Result] Peltzer K, Pengpid S. High prevalence of depressive symptoms in a national sample of adults in Indonesia: Childhood adversity, sociodemographic factors and health risk behaviour. Asian J Psychiatr. 2018 Mar;33:52-59. doi: 10.1016/j.ajp.2018.03.017. Epub 2018 Mar 7. PMID 29529418
- [Result] Rivera-Rivera Y, Vazquez-Santiago FJ, Albino E, Sanchez MD, Rivera-Amill V. Impact of Depression and Inflammation on the Progression of HIV Disease. J Clin Cell Immunol. 2016 Jun;7(3):423. doi: 10.4172/2155-9899.1000423. Epub 2016 Jun 3. PMID 27478681
- [Result] Anacker C. Adult hippocampal neurogenesis in depression: behavioral implications and regulation by the stress system. Curr Top Behav Neurosci. 2014;18:25-43. doi: 10.1007/7854_2014_275. PMID 24478038
- [Result] van Bodegom M, Homberg JR, Henckens MJAG. Modulation of the Hypothalamic-Pituitary-Adrenal Axis by Early Life Stress Exposure. Front Cell Neurosci. 2017 Apr 19;11:87. doi: 10.3389/fncel.2017.00087. eCollection 2017. PMID 28469557
- [Result] Islam MR, Islam MR, Ahmed I, Moktadir AA, Nahar Z, Islam MS, Shahid SFB, Islam SN, Islam MS, Hasnat A. Elevated serum levels of malondialdehyde and cortisol are associated with major depressive disorder: A case-control study. SAGE Open Med. 2018 May 9;6:2050312118773953. doi: 10.1177/2050312118773953. eCollection 2018. PMID 29770218
- [Result] Kambeitz JP, Howes OD. The serotonin transporter in depression: Meta-analysis of in vivo and post mortem findings and implications for understanding and treating depression. J Affect Disord. 2015 Nov 1;186:358-66. doi: 10.1016/j.jad.2015.07.034. Epub 2015 Jul 31. PMID 26281039
- [Result] Practice guideline for the treatment of patients with major depressive disorder (revision). American Psychiatric Association. Am J Psychiatry. 2000 Apr;157(4 Suppl):1-45. No abstract available. PMID 10767867
- [Result] Geurts DEM, Compen FR, Van Beek MHCT, Speckens AEM. The effectiveness of mindfulness-based cognitive therapy for major depressive disorder: evidence from routine outcome monitoring data. BJPsych Open. 2020 Nov 25;6(6):e144. doi: 10.1192/bjo.2020.118. PMID 33234183
- [Result] Worthington EL Jr, Hook JN, Davis DE, McDaniel MA. Religion and spirituality. J Clin Psychol. 2011 Feb;67(2):204-14. doi: 10.1002/jclp.20760. PMID 21108313
- [Result] Captari LE, Hook JN, Hoyt W, Davis DE, McElroy-Heltzel SE, Worthington EL Jr. Integrating clients' religion and spirituality within psychotherapy: A comprehensive meta-analysis. J Clin Psychol. 2018 Nov;74(11):1938-1951. doi: 10.1002/jclp.22681. Epub 2018 Sep 16. PMID 30221353
- [Result] Elkins GR, Barabasz AF, Council JR, Spiegel D. Advancing research and practice: the revised APA Division 30 definition of hypnosis. Int J Clin Exp Hypn. 2015;63(1):1-9. doi: 10.1080/00207144.2014.961870. PMID 25365125
- [Result] Alladin A. Evidence-based hypnotherapy for depression. Int J Clin Exp Hypn. 2010 Apr;58(2):165-85. doi: 10.1080/00207140903523194. PMID 20390689
- [Result] White L. Mindfulness in nursing: an evolutionary concept analysis. J Adv Nurs. 2014 Feb;70(2):282-94. doi: 10.1111/jan.12182. Epub 2013 Jun 16. PMID 23772683
- [Result] Valentine KE, Milling LS, Clark LJ, Moriarty CL. THE EFFICACY OF HYPNOSIS AS A TREATMENT FOR ANXIETY: A META-ANALYSIS. Int J Clin Exp Hypn. 2019 Jul-Sep;67(3):336-363. doi: 10.1080/00207144.2019.1613863. PMID 31251710
- [Result] Qin DD, Rizak J, Feng XL, Yang SC, Lu LB, Pan L, Yin Y, Hu XT. Prolonged secretion of cortisol as a possible mechanism underlying stress and depressive behaviour. Sci Rep. 2016 Jul 22;6:30187. doi: 10.1038/srep30187. PMID 27443987
- [Result] Garland EL, Hanley AW, Baker AK, Howard MO. Biobehavioral Mechanisms of Mindfulness as a Treatment for Chronic Stress: An RDoC Perspective. Chronic Stress (Thousand Oaks). 2017 Feb;1:2470547017711912. doi: 10.1177/2470547017711912. Epub 2017 Jun 22. PMID 28840198
- [Result] Milling LS, Valentine KE, McCarley HS, LoStimolo LM. A Meta-Analysis of Hypnotic Interventions for Depression Symptoms: High Hopes for Hypnosis? Am J Clin Hypn. 2019 Jan;61(3):227-243. doi: 10.1080/00029157.2018.1489777. PMID 34874235
- [Result] Yohn CN, Gergues MM, Samuels BA. The role of 5-HT receptors in depression. Mol Brain. 2017 Jun 24;10(1):28. doi: 10.1186/s13041-017-0306-y. PMID 28646910
- [Result] Jensen MP, Adachi T, Tome-Pires C, Lee J, Osman ZJ, Miro J. Mechanisms of hypnosis: toward the development of a biopsychosocial model. Int J Clin Exp Hypn. 2015;63(1):34-75. doi: 10.1080/00207144.2014.961875. PMID 25365127
- [Result] Marchand WR. Neural mechanisms of mindfulness and meditation: Evidence from neuroimaging studies. World J Radiol. 2014 Jul 28;6(7):471-9. doi: 10.4329/wjr.v6.i7.471. PMID 25071887
- [Result] Olendzki N, Elkins GR, Slonena E, Hung J, Rhodes JR. Mindful Hypnotherapy to Reduce Stress and Increase Mindfulness: A Randomized Controlled Pilot Study. Int J Clin Exp Hypn. 2020 Apr-Jun;68(2):151-166. doi: 10.1080/00207144.2020.1722028. PMID 32223617
- [Result] Elkins GR, Roberts RL, Simicich L. Mindful Self-Hypnosis for Self-Care: An Integrative Model and Illustrative Case Example. Am J Clin Hypn. 2018 Jul;61(1):45-56. doi: 10.1080/00029157.2018.1456896. PMID 29771220
- [Result] Otani A. Hypnosis and Mindfulness: The Twain Finally Meet. Am J Clin Hypn. 2016 Apr;58(4):383-98. doi: 10.1080/00029157.2015.1085364. PMID 27003487
- [Result] Doll A, Holzel BK, Mulej Bratec S, Boucard CC, Xie X, Wohlschlager AM, Sorg C. Mindful attention to breath regulates emotions via increased amygdala-prefrontal cortex connectivity. Neuroimage. 2016 Jul 1;134:305-313. doi: 10.1016/j.neuroimage.2016.03.041. Epub 2016 Mar 24. PMID 27033686